CLINICAL TRIAL: NCT02886494
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel, Phase II Study to Evaluate Efficacy and Safety of BAC in Patient With Alzheimer's Disease or Vascular Dementia
Brief Title: A Study to Evaluate Efficacy and Safety of BAC in Patient With Alzheimer's Disease or Vascular Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charsire Biotechnology Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BAC-02
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Results first posted 2021-07-19 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Alzheimer's Disease or Vascular Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- BAC treatment (Active Comparator): BAC, topical application on external nasal skin, scalp, and neck, 2 times daily, 30 g/day for 12 weeks
  Interventions: Drug: BAC treatment
- Matched vehicle (Placebo Comparator): Matched vehicle, topical application on external nasal skin, scalp, and neck, 2 times daily, 30 g/day for 12 weeks
  Interventions: Drug: Matched vehicle

INTERVENTIONS:
Drug: BAC treatment — BAC, topical application on external nasal skin, scalp, and neck, 2 times daily, 30 g/day for 12 weeks
  Other Names: CSTC1-BAC
  Arms: BAC treatment
Drug: Matched vehicle — BAC matched vehicle, topical application on external nasal skin, scalp, and neck, 2 times daily, 30 g/day for 12 weeks
  Other Names: Placebo control
  Arms: Matched vehicle

SUMMARY:
A Randomized, Double-Blind, Vehicle-Controlled, Parallel, Phase II Study to Evaluate Efficacy and Safety of BAC in Patient with Alzheimer's Disease or Vascular Dementia

DETAILED DESCRIPTION:
This study was designed as a randomized, double-blind, vehicle-controlled and parallel trial to evaluate the efficacy and safety of BAC in patients with Alzheimer's disease or vascular dementia. The investigation product, BAC, is a potential anti-inflammatory agent consisted of Multi-Glycan Complex (MGC) from the Soybean extract. It aims to reduce the neruoinflammation in the Alzhemimer's disease and vascular dementia.

In each study site, eligible patients were randomized and stratified to 1 of 2 dementia types (Alzheimer's disease and non-Alzheimer's disease) in 3:1 ratio to receive either one of topical application of BAC or BAC matched vehicle, topical application on external nasal skin, scalp, and neck, 2 times daily, 30 g/day.

The treatment duration for each patient was 12 weeks, which consisted of 6 visits located at Screening (within 2 weeks before Baseline visit), Baseline (Week 0), Weeks 2, 4, 8, and Week 12 (Final). During the treatment period, patients may continue to receive medications or treatments routinely used for Alzheimer's disease or vascular dementia except those prohibited under this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. With either gender aged at least 40 years old
2. With a diagnosis of one of the following disease i. Vascular dementia according to the NINDS-AIREN International Workshop criteria or ii. Alzheimer's disease according to the NIAAA criteria iii. "Mixed" dementia (possible Alzheimer's disease with cerebrovascular disease) according to the NIAAA criteria

   Note:
   1. NINDS-AIREN: National Institute of Neurological Disorders and Stroke and Association Internationale pour la Recherche et l'Enseignement en Neurosciences
   2. NIAAA: National Institute on Aging-Alzheimer's Association
3. With mild-to-moderate dementia (score of the Mini-Mental State Examination (MMSE) defined as between 10 to 24 and score of ADAS-Cog as at least 12)
4. Able to read, write, communicate, and understand cognitive testing instructions
5. Having a responsible caregiver who spends at least 4 hours daily with the patient. The caregiver will accompany the patient to all study visits, , supervise administration of study drug, and be able to assess the patient's condition
6. Patients and the responsible caregiver willing and able to provide written informed consent form

Exclusion Criteria:

1. With large vessel thrombosis (thrombotic stroke occurring in large arteries)
2. With radiological evidence of other brain disorders (subdural hematoma, post-traumatic / post-surgery)
3. With dementia caused by other brain diseases except Alzheimer's disease and vascular dementia (e.g. Parkinson's disease, demyelinated disease of the central nervous system, tumor, hydrocephalus, head injury, central nervous system infection including syphilis, acquired immune deficiency syndrome, etc.)
4. With clinical evidence of pulmonary, hepatic, gastrointestinal, metabolic, endocrine or other life threatening diseases judged by investigators not suitable to enter the study
5. With clinically unstable hypertension, diabetes mellitus, and cardiac disease for the last 3 months
6. Ever hospitalized for stroke or with acute coronary syndrome in the previous 3 months prior to screening
7. Drug or alcohol abuse within the previous 12 months of screening.
8. With one of the following abnormal laboratory parameters: hemoglobin < 10 mg/dL or platelet < 100*109/L; creatinine or total bilirubin more than 1.5 times the upper limit value; alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphates (ALP), γ-glutamyl transferase (γ-GT) more than 2 times the upper limit of normal, or thyroid-stimulating hormone (TSH) more than 2.5 times the upper limit value or less than the lower limit value of normal
9. With severe depression graded by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and Cornell Scale for Depression in Dementia (CSDD)
10. With any uncontrolled illness (including, but not limited to, any of the following: ongoing or active infection including hepatitis B, C, and HIV, active bleeding, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris or, cardiac arrhythmia) judged by the investigator that entering the trial may be detrimental to the patient
11. With known or suspected hypersensitivity to any ingredients of study product and vehicle
12. Pregnant or lactating or premenopausal with childbearing potential but not taking reliable contraceptive method(s) during the study period

    Note: Reliable contraceptive methods will consider as below:
    1. Established use of oral, injected or implanted hormonal methods of contraception > 3 months prior to baseline.
    2. Placement of an intrauterine device (IUD) or intrauterine system (IUS) > 3 months prior to baseline.
    3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
    4. Partner male sterilization (i.e., vasectomy) > 1 month of screening
13. Enrollment in any investigational drug trial within 4 weeks of screening visit
14. Experienced dosage increment of routinely use in drugs listed as follows within past three months before Screening visit

    1. medications/treatments for Alzheimer's disease or vascular dementia
    2. antipsychotic medications including but not limited to selective serotonin reuptake inhibitors (SSRIs), benzodiazepine (BZD)
    3. Vitamin B12
    4. drugs for thyroid disease
15. Current antiplatelet drug (antiaggregant) except dosage including but not limited to aspirin <= 100mg/day, clopidogrel <= 75mg/day, ticagrelor <= 180mg/day, dipyridamole <= 400mg/day
16. Caregivers who have psychotic symptoms, are imminently suicidal, have an unstable medical condition (e.g. recent heart attack, recent stroke, episodes of dizziness, fainting attacks) or significant orthopaedic problems.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Thein, Principal Investigator — Pacific Research Network
Locations (10):
- United States (10):
  - Clinical Research Consortium, Tempe, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - Pacific Research Network, LLC, San Diego, California
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - The Cognitive and Research Center of NJ, Springfield, New Jersey
  - Advanced Memory Research Institute of NJ, PC, Toms River, New Jersey
  - SPRI, Brooklyn, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Neurology Diagnostics, Inc., Dayton, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted in the United States. The study was open for recruitment in December 2016 and the first participant was successfully enrolled in January 2017.
Pre-assignment Details: The planned sample size was determined to be 45 versus 15 patients (3:1 ratio) for BAC treatment versus vehicle groups, 60 evaluable patients in total. To ensure the completion of 60 evaluable patients, around 75 patients were planned to be recruited. Actually, in this study, 80 eligible subjects were recruited and 59 evaluable subjects were achieved.
Groups:
- BAC Treatment: BAC, topically on external nasal skin, scalp, and neck, 30 g/day, 2 times daily for 12 weeks.
  Subjects were randomized 3:1 to receive double blind treatment of BAC or matched vehicle
- Matched Vehicle: BAC matched vehicle, topically on external nasal skin, scalp, and neck, 30 g/day, 2 times daily for 12 weeks
Period: Overall Study
Arm/Group | BAC Treatment | Matched Vehicle
Started | 60 | 20
Completed | 43 | 16
Not Completed | 17 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 12 | 3
Not completed — Protocol Violation | 4 | 1

BASELINE CHARACTERISTICS:
Population: [Not Specified]
Groups:
- Total: Total of all reporting groups
Arm/Group | BAC Treatment | Matched Vehicle | Total
Number analyzed (Participants) | 60 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (9.65) | 73.1 (9.19) | 73.2 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 11 | 52
  Male | 19 | 9 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Africa Americans | 5 | 2 | 7
  Race: Caucasians | 54 | 17 | 71
  Race: Hispanic | 1 | 0 | 1
  Race: Hispanic Native American | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 20 | 80
Dementia history [Count of Participants; unit: Participants]
  Alzheimer's Disease | 42 | 13 | 55
  Mixed Dementia | 11 | 6 | 17
  Vascular Dementia | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Alzheimer Disease Assessment Scale-cognitive (ADAS-cog) Score at Week 12 Visit Compared to Baseline
Description: The Alzheimer's Disease Assessment Scale- Cognitive (ADAS-Cog) Subscale test is the standard assessment tool and one of the most popular cognitive testing instrument in clinical trials. It is designed to assess various cognitive abilities such as those associated with memory, language and praxis. It consists of 11 parts: 1. Word Recall Task; 2. Naming Task; 3: Commands; 4: Constructional Praxis; 5. Ideational Praxis; 6. Orientation; 7. Word Recognition Task; 8. Language; 9. Comprehension of Spoken Language; 10. Word Finding Difficulty; and 11. Remembering Test Instructions. Scores range from 0 to 70 with lower scores indicating lesser severity. ADAS-Cog was measured at Screening, Randomization/Baseline, Week 4, Week 8 and Week 12.
Time Frame: Week 12
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BAC Treatment: BAC, topically on external nasal skin, scalp, and neck, 30 g/day, 2 times daily for 12 weeks
Arm/Group | BAC Treatment | Matched Vehicle
Number analyzed (Participants) | 44 | 16
score on a scale | -0.05 (5.726) | -2.25 (4.973)

2. Secondary Outcome: Change in ADAS-cog Score at All Post Treatment Visits (Except Week 12 Visit) Compared to Baseline
Description: as for outcome 1
Time Frame: Week 4, 8
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BAC Treatment Arm: BAC, topically on external nasal skin, scalp, and neck, 30 g/day, 2 times daily for 12 weeks
- BAC Matched Vehicle: BAC matched vehicle, topically on external nasal skin, scalp, and neck, 30 g/day, 2 times daily for 12 weeks
Arm/Group | BAC Treatment Arm | BAC Matched Vehicle
Number analyzed (Participants) | 60 | 20
score on a scale
  Week 4 - Baseline: number analyzed (Participants) | 51 | 18
  Week 4 - Baseline | -0.51 (4.096) | -2.33 (4.393)
  Week 8 - Baseline: number analyzed (Participants) | 48 | 17
  Week 8 - Baseline | -0.79 (4.177) | -2.06 (5.068)

3. Secondary Outcome: Clinician's Interview Based Impression of Change-Plus Caregiver Input (CIBIC-plus) Score at All Post Treatment Visits
Description: This is a global measure of detectable change in cognition, function and behavior. The format for CIBIS/CIBIC-Plus consists of the assessment of an independent clinician based on observation of the patient at an interview, and information provided by the caregiver. The clinician's assessing severity at baseline and overall impression for assessing severity of the global change in disease severity, compared with baseline, is rated. The CIBIS/CIBIC plus examined general, cognitive, and behavioral function and activities of daily living on a 7-point categorical rating scale, ranging from a score of 0 indicating "Not assessed", to a score of 7 indicating "Among the most extremely ill patients" for CIBIS and ranging from 1 indicating "Very much improved", to a score of 7 indicating "Marked worsening", and with a score of 4 indicating "no change" for CIBIC-Plus. CIBIS was measured at Randomization visit and CIBIC-Plus was measured at Week 4, Week 8, and Week 12.
Time Frame: Week 4, 8, 12
Population: All randomized patients who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Matched Vehicle: Matched vehicle, topically on external nasal skin, scalp, and neck, 30 g/day, 2 times daily for 12 weeks
Arm/Group | BAC Treatment | Matched Vehicle
Number analyzed (Participants) | 60 | 20
Participants
  Week 4: number analyzed (Participants) | 51 | 18
  Week 4: 1. Very much improved | 0 | 0
  Week 4: 2. Much improved | 1 | 1
  Week 4: 3. Minimal improved | 6 | 3
  Week 4: 4. No change | 41 | 10
  Week 4: 5. Minimal worsening | 3 | 4
  Week 4: 6. Moderate worsening | 0 | 0
  Week 8: number analyzed (Participants) | 48 | 17
  Week 8: 1. Very much improved | 0 | 0
  Week 8: 2. Much improved | 1 | 1
  Week 8: 3. Minimal improved | 2 | 1
  Week 8: 4. No change | 36 | 13
  Week 8: 5. Minimal worsening | 8 | 2
  Week 8: 6. Moderate worsening | 1 | 0
  Week 12: number analyzed (Participants) | 44 | 16
  Week 12: 1. Very much improved | 1 | 0
  Week 12: 2. Much improved | 1 | 2
  Week 12: 3. Minimal improved | 2 | 0
  Week 12: 4. No change | 33 | 11
  Week 12: 5. Minimal worsening | 5 | 3
  Week 12: 6. Moderate worsening | 2 | 0

4. Secondary Outcome: Change in Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Score at All Post Treatment Visits Compared to Baseline
Description: An inventory of informant based items to assess activities of daily living and instrumental activities of daily living, i.e. functional performance, of Alzheimer's disease (AD). It consists of 23-item inventory of ADL, rated based on extent of assistance the patient requires (independently, with supervision, with physical help): 0 (total independence in performing an activity) to 4 (total inability to act independently). Each question varies in the number of options to choose. Total score range: 0 to 78; higher scores indicate less functional impairment. ADL will be measured at Randomization/Baseline, Week 4, Week 8, and Week 12.
Time Frame: Week 4, 8, 12
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BAC Treatment | Matched Vehicle
Number analyzed (Participants) | 60 | 20
score on a scale
  Week 4 - Baseline: number analyzed (Participants) | 51 | 18
  Week 4 - Baseline | -0.71 (3.613) | 1.17 (4.618)
  Week 8 - Baseline: number analyzed (Participants) | 48 | 17
  Week 8 - Baseline | 0.08 (3.188) | 0.53 (6.084)
  Week 12 - Baseline: number analyzed (Participants) | 44 | 16
  Week 12 - Baseline | 0.23 (3.241) | 1.75 (5.422)

5. Secondary Outcome: Change in Mini-Mental State Examination (MMSE) Score at All Post Treatment Visits Compared to Baseline
Description: This is a multi-item instrument that examines orientation, registration, attention, calculation, recall, visuospatial abilities and language. The score ranges from 0 to 30, with higher scores indicating better cognitive function. MMSE was measured at Screening, Randomization/Baseline, Week 4, Week 8, and Week 12.
Time Frame: Week 4, 8, 12
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BAC Treatment | Matched Vehicle
Number analyzed (Participants) | 60 | 20
score on a scale
  Week 4 - Baseline: number analyzed (Participants) | 51 | 18
  Week 4 - Baseline | 0.61 (2.089) | 0.17 (2.431)
  Week 8 - Baseline: number analyzed (Participants) | 48 | 17
  Week 8 - Baseline | 0.25 (1.732) | 1.35 (2.691)
  Week 12 - Baseline: number analyzed (Participants) | 44 | 16
  Week 12 - Baseline | 0.43 (2.182) | 0.56 (2.476)

6. Secondary Outcome: Change in Neuropsychiatric Inventory (NPI) Score at All Post Treatment Visits Compared to Baseline: NPI-10 Frequency × Severity
Description: The NPI is the behavior instrument most widely used in clinical trials of anti-dementia agents. The NPI uses a screening strategy to minimize administration time, examining and scoring only those behavioral domains with positive responses to screening questions. Both the frequency and the severity of each behavior are determined. Information for the NPI is obtained from a caregiver familiar with the patient's behavior. The NPI assesses 10 behavioral domains (10-item NPI, section A~J) common in dementia. Each NPI domain is scored by the caregiver based on a standardized interview administered by the clinician. Frequency is scored from 1 (occasionally) to 4 (very frequently) and severity is rated from 1 (mild) to 3 (severe). The score for each domain is frequency multiplied by severity. Therefore, the score ranges from 1 to 12 with higher scores indicate worse condition. NPI was measured at Randomization/Baseline, Week 4, Week 8, and Week 12.
Time Frame: Week 4, 8, 12
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BAC Treatment | Matched Vehicle
Number analyzed (Participants) | 60 | 20
score on a scale
  Week 4 - Baseline: number analyzed (Participants) | 51 | 18
  Week 4 - Baseline | -0.37 (8.607) | -2.28 (6.952)
  Week 8 - Baseline: number analyzed (Participants) | 48 | 17
  Week 8 - Baseline | -0.75 (4.024) | -2.76 (6.250)
  Week 12 - Baseline: number analyzed (Participants) | 44 | 16
  Week 12 - Baseline | -1.48 (6.550) | -3.13 (6.672)

7. Secondary Outcome: Change in Neuropsychiatric Inventory (NPI) Score at All Post Treatment Visits Compared to Baseline: NPI-10 Caregiver Distress Score
Description: The NPI is the behavior instrument most widely used in clinical trials of anti-dementia agents. The NPI uses a screening strategy to minimize administration time, examining and scoring only those behavioral domains with positive responses to screening questions. Both the frequency and the severity of each behavior are determined. Information for the NPI is obtained from a caregiver familiar with the patient's behavior. The NPI assesses 10 behavioral domains (10-item NPI) common in dementia. Each NPI domain is scored by the caregiver based on a standardized interview administered by the clinician. NPI-10 Caregiver Distress score is scored for associated caregiver distress from 0 (no distress) to 5 (very severe or extreme). Higher scores indicate greater distress. NPI was measured at Randomization/Baseline, Week 4, Week 8, and Week 12.
Time Frame: Week 4, 8, 12
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BAC Treatment | Matched Vehicle
Number analyzed (Participants) | 60 | 20
score on a scale
  Week 4 - Baseline: number analyzed (Participants) | 51 | 18
  Week 4 - Baseline | -0.02 (2.839) | -1.94 (4.094)
  Week 8 - Baseline: number analyzed (Participants) | 48 | 17
  Week 8 - Baseline | -0.52 (1.902) | -2.06 (4.451)
  Week 12 - Baseline: number analyzed (Participants) | 44 | 16
  Week 12 - Baseline | -0.91 (2.595) | -2.25 (4.740)

8. Secondary Outcome: Change in Neuropsychiatric Inventory (NPI) Score at All Post Treatment Visits Compared to Baseline: NPI-12 Frequency × Severity Score
Description: The NPI is the behavior instrument most widely used in clinical trials of anti-dementia agents. The NPI uses a screening strategy to minimize administration time, examining and scoring only those behavioral domains with positive responses to screening questions. Both the frequency and the severity of each behavior are determined. Information for the NPI is obtained from a caregiver familiar with the patient's behavior. The NPI assesses 12 behavioral domains (12-item NPI) common in dementia. Each NPI domain is scored by the caregiver based on a standardized interview administered by the clinician. Frequency is scored from 1 (occasionally) to 4 (very frequently) and severity is rated from 1 (mild) to 3 (severe). The score for each domain is frequency multiplied by severity. Therefore, the score ranges from 1 to 12 with higher scores indicate worse condition. NPI was measured at Randomization/Baseline, Week 4, Week 8, and Week 12.
Time Frame: Week 4, 8, 12
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BAC Treatment | Matched Vehicle
Number analyzed (Participants) | 60 | 20
score on a scale
  Week 4 - Baseline: number analyzed (Participants) | 51 | 18
  Week 4 - Baseline | -0.61 (9.944) | -3.89 (9.074)
  Week 8 - Baseline: number analyzed (Participants) | 48 | 17
  Week 8 - Baseline | -1.29 (6.348) | -4.76 (9.437)
  Week 12 - Baseline: number analyzed (Participants) | 44 | 16
  Week 12 - Baseline | -1.80 (8.582) | -5.50 (10.047)

9. Secondary Outcome: Change in Neuropsychiatric Inventory (NPI) Score at All Post Treatment Visits Compared to Baseline: NPI-12 Caregiver Distress Score
Description: The NPI is the behavior instrument most widely used in clinical trials of anti-dementia agents. The NPI uses a screening strategy to minimize administration time, examining and scoring only those behavioral domains with positive responses to screening questions. Both the frequency and the severity of each behavior are determined. Information for the NPI is obtained from a caregiver familiar with the patient's behavior. The NPI assesses 12 behavioral domains (12-item NPI) common in dementia. Each NPI domain is scored by the caregiver based on a standardized interview administered by the clinician. NPI-12 Caregiver Distress score is scored for associated caregiver distress from 0 (no distress) to 5 (very severe or extreme). Higher scores indicate greater distress. NPI was measured at Randomization/Baseline, Week 4, Week 8, and Week 12.
Time Frame: Week 4, 8, 12
Population: All randomized patients who have received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BAC Treatment | Matched Vehicle
Number analyzed (Participants) | 60 | 20
score on a scale
  Week 4 - Baseline: number analyzed (Participants) | 51 | 18
  Week 4 - Baseline | -0.02 (3.010) | -2.56 (5.193)
  Week 8 - Baseline: number analyzed (Participants) | 48 | 17
  Week 8 - Baseline | -0.67 (2.291) | -2.76 (5.815)
  Week 12 - Baseline: number analyzed (Participants) | 44 | 16
  Week 12 - Baseline | -0.93 (2.840) | -3.13 (6.174)

10. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a study medication and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a study medication, whether or not related to the study medication. Laboratory abnormalities should not be recorded as AEs unless determined to be clinically significant by the Investigator. The number of participants with adverse events within the BAC and placebo groups was determined.
Time Frame: AEs were reported through the study completion (up to 12 weeks)
Population: All randomized patients who have received at least one dose study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | BAC Treatment | Matched Vehicle
Number analyzed (Participants) | 60 | 20
Participants | 20 | 7

11. Post Hoc Outcome: "Responder" Analysis of MMSE Score at All Post Treatment Visits Compared to Baseline, on All Subjects Not Receiving Any Dementia Medication (Naïve)
Description: This is a multi-item instrument that examines orientation, registration, attention, calculation, recall, visuospatial abilities and language. The maximum score is 30, with higher scores indicating better cognitive function. ).
  "Responder" analysis consist of two steps. (1) The baseline MMSE score is deducted from the post-treatment visit MMSE score; (2) the minus baseline score in step 1 is being dichotomized into two binary variable of either "responder" or "non-responder". Patients who make progress or remain unchanged on the cognitive test compared to baseline are considered as "responders", whereas patients who have deterioration on the cognitive test compared to baseline are considered as "non-responders".
Time Frame: Week 4, 8, 12
Population: All randomized patients who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | BAC Treatment | Matched Vehicle
Number analyzed (Participants) | 60 | 20
Participants
  Week 4 - baseline: number analyzed (Participants) | 17 | 8
  Week 4 - baseline | 13 | 5
  Week 8 - baseline: number analyzed (Participants) | 15 | 8
  Week 8 - baseline | 12 | 6
  Week 12 - baseline: number analyzed (Participants) | 14 | 7
  Week 12 - baseline | 12 | 5

12. Post Hoc Outcome: "Responder" Analysis of ADAS-cog Score at All Post Treatment Visits Compared to Baseline, on All Subjects Not Receiving Any Dementia Medication (Naïve)
Description: The ADAS-Cog Subscale test is the standard assessment tool and one of the most popular cognitive testing instrument in clinical trials. It is designed to assess various cognitive abilities such as those associated with memory, language and praxis. Scores range from 0 to 70 with lower scores indicating lesser severity.
  "Responder" analysis consist of two steps. (1) The baseline ADAS-cog score score is deducted from the post-treatment visit ADAS-cog score; (2) the minus baseline score in step 1 is being dichotomized into two binary variable of either "responder" or "non-responder". Patients who make progress or remain unchanged on the cognitive test are considered as "responders", whereas patients who have deterioration on the cognitive test are considered as "non-responders".
Time Frame: Week 4, 8, and 12
Population: All randomized patients who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | BAC Treatment | Matched Vehicle
Number analyzed (Participants) | 60 | 20
Participants
  Week 4 - Baseline: number analyzed (Participants) | 17 | 8
  Week 4 - Baseline | 13 | 7
  Week 8 - Baseline: number analyzed (Participants) | 15 | 8
  Week 8 - Baseline | 10 | 6
  Week 12 - Baseline: number analyzed (Participants) | 14 | 7
  Week 12 - Baseline | 11 | 4

ADVERSE EVENTS:
Time Frame: AE data was collected from Screening visit to Final visit (up to 12 weeks)
Description: All enrolled subjects were used for the analysis of AE and SAE.
Arm/Group | BAC Treatment | Matched Vehicle
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/20
Other Adverse Events (participants affected / at risk) | 6/60 | 7/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BAC Treatment (N=60) | Matched Vehicle (N=20)
Nasopharyngitis (Infections and infestations) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 2
Somnolence (Nervous system disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT02886494/Prot_SAP_000.pdf